CLINICAL TRIAL: NCT01666184
Title: Biomarkers Study in Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Chang Gung Memorial Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Mackay Memorial Hospital (Other); Taichung Veterans General Hospital (Other); National Cheng-Kung University Hospital (Other); Kaohsiung Veterans General Hospital. (Other); Kaohsiung Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: T3212
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Biomarkers Study in Pancreatic Cancer
Keywords: Biomarkers study

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The specimen and clinical information will be collected and delivered to the laboratory of Dr. Hui-Ju Ch'ang over NICR, NHRI, Tainan .
Oversight: Data Monitoring Committee: No

SUMMARY:
Study Design:

Patients are eligible if (1) enrolled to TCOG 3207(2) received surgery or biopsy for pancreatic cancer; (3) willing to sign informed consent.

The pancreatic tumor, tissue specimen and blood sample before or after treatment will be collected from department of pathology, surgery or diagnostic medicine.

DETAILED DESCRIPTION:
We expect to collect tissue samples from 270 pancreatic cancer patients of any stages. Since the enrollment criteria are not limited to new patients, we expect to enroll 67 patients a year. The patient enrollment will be completed in 4 years. Clinical follow-up will be completed in another one year. Data analysis and correlation study may be finished in the end of 5th year of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients enrolled to TCOG 3207 study: A Randomized Phase III Study of Adjuvant Gemcitabine versus Gemcitabine Plus Concurrent Chemoradiation in Pancreatic Cancer Underwent Curative Intent (R0 / R1) Resection.
2. Patients who were not eligible for TCOG 3207 study but received surgery or biopsy for pancreatic cancer.
3. Patients have to sign informed consent for tissue specimen collection, according to the regulation of DOH.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We expect to collect tissue samples from 270 pancreatic cancer patients of resectable pancreatic cancer. Since the enrollment criteria are not limited to new patients, we expect to enroll 67 patients a year. The patient enrollment will be completed in 4 years. Clinical follow-up will be completed in another one year. Data analysis and correlation study may be finished in the end of 5th year of this study.
Sampling Method: Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2012-09; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Ming Shyr, M.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan; Tsann-Long Hwang, M.D., Principal Investigator — Chang Gung Memorial Hospital; Ruey-Kuen Hsieh, M.D., Principal Investigator — Mackay Memorial Hospital Taipei, Taiwan

REFERENCES:
- [Derived] Tsai YC, Chen SL, Peng SL, Tsai YL, Chang ZM, Chang VH, Ch'ang HJ. Upregulating sirtuin 6 ameliorates glycolysis, EMT and distant metastasis of pancreatic adenocarcinoma with kruppel-like factor 10 deficiency. Exp Mol Med. 2021 Oct;53(10):1623-1635. doi: 10.1038/s12276-021-00687-8. Epub 2021 Oct 26. PMID 34702956